CLINICAL TRIAL: NCT04657354
Title: Return to Work After Early Intervention for Lumbar Disc Herniation Versus Usual Care
Acronym: WILD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough patients
Sponsor: Spine Centre of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/34764
Record Dates: First submitted 2020-11-02; First posted 2020-12-08 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Herniated Disk Lumbar
Keywords: rct; wild; Return to work; sick leave; sciatica; lumbar pain; Radiculopathy; Spine; Quality of life; Herniated lumbar disc
MeSH Terms: conditions — Sciatica; Low Back Pain; Radiculopathy | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast track (Active Comparator): Study subjects in Fast Track arm will get an MRI done on the same day. If the MRI shows concordant findings of herniated disc, the subject will be referred to a spine surgeon to be seen within one week. If the surgeon and subject decide on discectomy, the surgery is scheduled within the same week. Total timespan from first interview to surgery will be no longer than 2 weeks.
  Interventions: Procedure: Assessment
- Usual care (No Intervention): Study subjects in Usual Care will be treated following the Danish National Guidelines in which a conservative approach for the first 4-6 weeks with focus on pain relief by pain-relief medication, exercises and encouragement to resume normal activities as much as possible. Patients in this arm will be scheduled 2 and 4 week follow-up appointments as per national guidelines.
  If the symptoms have not resolved after this period, then a referral to a multidisciplinary spine care department is made. However, if symptoms are still present at 8-12 weeks first then a referral for a spine surgeon assesment can be done.

INTERVENTIONS:
Procedure: Assessment — Early surgical assessment
  Arms: Fast track

SUMMARY:
The most common cause of low back pain with radiculopathy among the working population is a Lumbar Disc Herniation (LDH). In general, the natural history of sciatica is favourable with spontaneous remission. For the subgroup with more severe symptoms that do not resolve the vocational prognosis is unfavourable in more than 1/3 of the patients. Factors negatively affecting return to work were unskilled labour and less than 40 weeks of employment.

Other than poorer prognosis for patients undergoing discectomy six months or later after the onset of symptoms, there is no consensus on the timing of discectomy. National guidelines in Denmark recommend referral to a spine surgeon if the patient's symptoms have not resolved within 8-12 weeks. However, recent studies have shown that duration of sick leave is associated with poorer clinical outcomes and lower return to work rates.

The purpose of this study is to establish if early surgical evaluation of patients with symptomatic LDH can improve return to work rates. A secondary purpose is to analyse the socioeconomic benefits or costs of an earlier surgical evaluation.

This is a randomized controlled study of two parallel groups of patients who contact their general practitioner for pain relief due to LDH and have been on a minimum of 2 weeks of paid leave. The patients will be randomised to either fast track surgical evaluation or usual care. After informed consent, the subjects will be followed for a period of 12 months.

There are ethical considerations to address including the potential risk of performing surgery if the patient's symptoms could have resolved spontaneously. On the other hand, delayed discectomy could increase the risks of developing chronic pain and loss of work. Thus, the intervention being studied is early referral to a spine surgeon and not discectomy per se. This allows the subject to make a preference-based decision with the surgeon to have a discectomy or not.

DETAILED DESCRIPTION:
Design The study design will be a randomized parallel group prospective study of patients from the region of Southern Denmark and the region Zealand with sciatica due to LDH randomized to either early surgical evaluation or usual care as per recommendations from the Danish National Health Board

Study population Study subjects are identified from the patient population in the region of Southern Denmark and the Region of Zealand clinically diagnosed with LDH by their general practitioner.

Randomisation procedure Eligible patients are randomised into one of two arms, usual care or fast track surgical evaluation with a 1:1 Block sealed envelope randomisation used. A randomized block design, stratified by the two surgical sites, is used to ensure equal distribution of the two treatment arms in regions. The randomisation procedure is concealed and administered by the primary investigator. Randomisation is performed after the patient has signed the informed consent form. The result of the randomisation is documented in the subjects' trial record.

Study Arms:

Subject withdrawal If a subject develops a clinically significant medical or surgical condition that in the opinion of the investigator could impact the patient's ability to successfully complete the trial or otherwise interfere with outcomes, the subject will be withdrawn.

If the patient during the trial or follow-up period receives other medical or invasive intervention that in the opinion of the investigator could impact on the patient's ability to successfully complete the trial or otherwise interfere with outcomes, the subject will be withdrawn,

These subjects will not be included in the final analysis

Patient course In Denmark the General Practioners' (GP's) are organised in clusters to ensure a uniform quality of treatment. The study will be presented to all pre-existing GP-clusters in the two participating regions at a GP-cluster meeting prior to the study by investigator. Individual written consent from the GP to participate is obtained at the meeting. All GP's not present will be identified and contacted individually to obtain written consent. All participating GP's are informed and consent that all study subjects will, for the duration of the study, be seen and treated by the investigator GP regarding their LDH, to include all consultations, scripts, off work certificates, referrals etc. for as long as the patient is part of the study. All patient encounters will be documented, and relevant information given to respective GP's ongoing. Two laminated coloured A4 posters are distributed to each GP, one for the GP and one for reception with trial name, screening criteria and investigators phone number and e-mail.

Both the GP's who participate and don't participate in the study are recorded. All patients that meet screening criteria are asked if investigator can contact them by phone. Investigator then calls the patient to assess inclusion and exclusion criteria. If study subject is found eligible then they will be thoroughly informed of the study and informed consent is obtained per mail and an appointment for clinic visit with the Principal Investigator is scheduled within one week is given. Information and inclusion of participants will be conducted in accordance with the guidelines of the Health Research Ethics Committee System in Denmark, from which approval will be sought.

During the first interview and examination, all study subjects' complete questionnaires as per Table 1.

Study subjects in Usual Care will be treated following the Danish National Guidelines; get relevant prescriptions, certificates, x-ray and physio/chiropractor referral as per standard recommendations Study subjects in Fast Track arm will get an MRI done on the same day. All MRIS will be performed and read at Middelfart Sygehus or Zealand University Hospital. If the MRI shows concordant findings of herniated disc, the subject will be referred to a spine surgeon to be seen within one week.

The surgeon will assess the patient and ensure the magnetic resonance image (MRI) demonstrates a lumbar disc herniation, with the level and side corresponding with clinical symptoms such as lower extremity radicular pain and/or affection of neurological function. The subject and the surgeon will discuss the benefits and risks of a discectomy with the subject. A decision regarding discectomy will be made taking into consideration the subject's preference. If the surgeon and subject decide on discectomy, the surgery is scheduled within the same week. Total timespan from first interview to surgery will be no longer than 2 weeks.

All discectomies for subjects in Fast Track arm will be performed at one of three Spine Surgery Centres, Middelfart Sygehus, Odense Universitets Hospital (OUH) or Department of Orthopaedic Surgery, Zealand University Hospital, Køge. Depending on the surgeon's preference, the surgical techniques will vary between open discectomy with or without the use of microscope and tubular-discectomy.

Discectomies for subjects in Usual Care will be performed by a qualified spine surgeon but not necessary at one of the three centres.

All patients irrespectively to study arm and treatment site are scheduled to standard post-operative out-patient program with clinic visits as all Danish patients are legally entitled to a free course of rehabilitation in the municipal centers. Rehabilitation programs typically last 8-10 weeks and consist of either team or individual training 1-2 times weekly combined with home exercises (13) Study subjects in both arms will be mailed questionnaires as per table 1 and a SMS text reminder 3 days later if reply haven been recorded. This will be handled automatically by RedCap. If still no reply is recorded, then investigator will phone the study subject 7 days post mail.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed by their GP with LDH
* Sick leave due to LDH
* Duration of sick leave less 6 weeks.
* Age >= 18
* Able to understand and read Danish
* Informed consent

Exclusion Criteria:

* History of previous spine surgery or spinal fracture
* History of lumbar radiation therapy
* Current malignant disease or chemotherapy
* Current pregnancy or breast-feeding
* Diagnosis of significant psychiatric disorder
* Contra-indication for spinal surgery or rehabilitation
* Patients that are not eligible to have an MRI scan
* Presence of neurologic deficit requiring urgent decompressive spinal surgery

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Working age
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Return to work | 12 months
  Self-reported work status. Return to work status one year after entry.

SECONDARY OUTCOMES:
Socioeconomic costs | 12 months
  The Incremental Cost-Effectiveness Ratios (ICER) will be calculated as the difference in cost between the two groups divided by the difference in QALYs gained or lost.
Patient reported outcome | 12 months
  To evaluate pain we will use VAS scale used measure from 0-100 where 0 is no pain and 100 is most pain.
Surgical rates | 12 months
  To measure surgical rates we use the Scandinavian national spine registre where all surgical procedures are recorded. Study subjects will be grouped within 2 weeks intervals defined from the time of pain onset to performed surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ankjaer, MD, Principal Investigator — Spine centre Middelfart University of Southerne Denmark

IPD SHARING:
Plan to Share IPD: No
It is the intention to publish the results, whether positive or negative, in relevant international high impact journals.